CLINICAL TRIAL: NCT01967563
Title: Effect of a Eucaloric Ketogenic Diet on Energy Expenditure: A Pilot Study
Brief Title: Study of the Effect of a Very-Low-Carbohydrate Diet on Energy Expenditure
Status: Terminated | Type: Observational
Why Stopped: PI is no longer at NIH
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Pennington Biological Research Center (Unknown); Translational Research Institute for Metabolism and Diabetes (Unknown); Columbia University, New York, NY (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130212; 13-DK-0212
Record Dates: First submitted 2013-10-22; First posted 2013-10-23 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Appetite; Healthy Volunteers
Keywords: Energy Expenditure; Obesity; Carbohydrate; Fat; Ketones; Natural History
MeSH Terms: conditions — Obesity; Platelet Glycoprotein IV Deficiency; Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- overweight and class I obese adult male volunteers: Adult Male Subjects will be recruited to determine the effects on energy expenditure of transitioning from an energy-and macronutrient-balanced standard baseline diet to a eucaloric ketogenic diet

SUMMARY:
Background:

- Popular weight loss plans often restrict carbohydrates or fat. Research shows that very-low-carbohydrate (ketogenic) diets lead to greater weight loss than low-fat diets. Researchers want to know if eating fewer carbohydrates changes the number of calories the body uses. They also want to know how a ketogenic diet affects hunger, hormones, and food preferences.

Objectives:

- To better understand how the body responds to different diets.

Eligibility:

- Men 18 to 50 years old who are healthy but overweight.

Design:

* Participants will have 3 screening visits:

  1. Medical history, physical exam, blood test, and EKG. They will eat during the visit.
  2. For the week before the visit, participants will wear physical activity monitors daily. They will record everything they eat and sample the special diet. At the visit, they will receive an EKG and heart rate test while biking for 30 minutes.
  3. For the week before the visit, participants will wear the physical activity monitors. They will eat all their meals from the special diet that will be provided. At the visit, they will answer questions and bike for 60 minutes.
* After screening, for 1 week, participants will visit the clinic daily to receive that day s food. They will not eat or drink anything else except water.
* Then participants will stay at the clinic for 8 weeks. They cannot leave but can have visitors. Participants will wear physical activity monitors, bike daily, and follow different diets. Tests will be given daily, and may include weighing, X-rays, and blood and urine tests. They will spend several days in a monitored room to test oxygen and carbon dioxide.

DETAILED DESCRIPTION:
Popular weight loss strategies often prescribe targeted reduction of dietary carbohydrate or fat. Recent clinical trials in obese subjects have found that low-carbohydrate diets result in greater weight loss compared with low-fat diets on a time scale of months when diet adherence was likely the highest. One hypothesis regarding the mechanism of improved weight loss with low carbohydrate diets is that such diets significantly modify the body s hormonal milieu to influence metabolic regulation and energy expenditure. Low-carbohydrate diets may thereby offer a metabolic advantage over low fat diets. In addition, low-carbohydrate diets may also decrease hunger or increase satiety compared to low-fat diets.

Determining the mechanism whereby one diet leads to greater weight loss than another is hampered by the inability to accurately measure food intake or physical activity in an outpatient setting. Thus, an inpatient feeding study lasting many weeks is required to accurately measure energy balance differences between isocaloric diets that differ in macronutrient composition. In this pilot multicenter cross-over study in 16 overweight and class I obese men, we will measure changes in energy expenditure in response to 4 weeks of inpatient feeding of a eucaloric, very low carbohydrate, ketogenic diet (5% Carbohydrate, 15% Protein, 80% Fat) immediately following an inpatient period of at least 4 weeks of consuming an energy balanced standard American diet (50% Carbohydrate, 15 % Protein, 35% Fat).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-50 years, male
* Weight stable (< 5 % over past 6 months)
* Current stable weight no more than 8% below lifetime maximum weight
* Body mass index (BMI) greater than or equal to 25 kg/m(2) but less than 35 kg/m(2), with each study site recruiting an equal number of subjects from the overweight range of 25 kg/m(2) less than or equal to BMI < 30 kg/m(2) and from the class I obese range of 30 kg/m(2) less than or equal to BMI < 35 kg/m(2)
* Otherwise healthy, as determined by medical history and laboratory tests
* Able to complete daily bouts of stationary cycling at a moderate rate and intensity
* Written informed consent
* Willing to eat all the food provided in the study
* Willing to continue consistently their habitual caffeine intake

EXCLUSION CRITERIA:

* BMI < 25 kg/m(2) or greater than or equal to 35 kg/m(2)
* Blood pressure > 140/90 mm Hg
* Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, diabetes, thyroid disease)
* Taking any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, asthma medication, blood pressure medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
* Hematocrit < 40%
* Participating in a regular exercise program (> 2h/week of vigorous activity)
* Dietary carbohydrate less than 30% or greater than 65% of total calories as determined by food frequency questionnaire
* Caffeine consumption > 300 mg/day
* Regular use of alcohol (> 2 drinks per day), tobacco (smoking or chewing) amphetamines, cocaine, heroin, or marijuana over past 6 months
* Past or present history of eating disorder (including binge eating) or psychiatric disease, including claustrophobia since part of the protocol will involve being confined to a small room for whole-body indirect calorimetry
* Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, multiple food allergies)
* Volunteers unwilling or unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will study the magnitude and variability of energy expenditure changes in response to a eucaloric ketogenic diet subsequent to a standard energy- and macronutrient-balanced diet in overweight and class I obese adult male volunteers
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
To determine 24hr energy expenditure, respiratory quotient, and sleeping energy expenditure following a 4-week eucaloric ketogenic diet as compared to 4 weeks of consuming an energy-balanced standard diet. | 1 year
  the subjects will spend the 4th, 5th, 11th, 12th, 18th, 19th, 25th and 26th days of Stages 2 & 3 in the metabolic chamber to measure 24-hour energy expenditure and sleeping energy expenditure. The energy expenditure calculations will be corrected for urinary ketone excretion since approximately 0.33 L of O2 is consumed for every gram of ketone excreted in the urine.

SECONDARY OUTCOMES:
To investigate changes in body composition and appetitive behaviors such as hunger, satiety, food impulsivity, and food liking & wanting during a 4-week eucaloric ketogenic diet as compared to 4 weeks of consuming an energy-balanced stan... | 7 days(outpatient) plus 8 weeks( inpatient)
  hunger and satiety assessments will be completed multiple times each day, and ad libitum meal tests and appetitive computer tasks (delay discounting, liking & wanting, go/no-go, food choice) will be performed during the latter periods of Stages 2 & 3.
To determine body weight and body composition following a 4-week eucaloric ketogenic diet as compared to 4 weeks of consuming an energy-balanced standard diet. | 7 days (outpatient) plus 8 weeks (inpatient)
  measurement of body composition by DXA, isotope dilution, and air-displacement plethysmography (BodPod) will be performed on the 15th and 28th days of Stages 2 & 3. Measurement of total body water by administering deuterium oxide will be performed on the 28th day of Stages 2 & 3. Body weight will be measured daily.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Rosenbaum M, Hall KD, Guo J, Ravussin E, Mayer LS, Reitman ML, Smith SR, Walsh BT, Leibel RL. Glucose and Lipid Homeostasis and Inflammation in Humans Following an Isocaloric Ketogenic Diet. Obesity (Silver Spring). 2019 Jun;27(6):971-981. doi: 10.1002/oby.22468. Epub 2019 May 8. PMID 31067015
- [Derived] Hall KD, Guo J, Chen KY, Leibel RL, Reitman ML, Rosenbaum M, Smith SR, Ravussin E. Methodologic considerations for measuring energy expenditure differences between diets varying in carbohydrate using the doubly labeled water method. Am J Clin Nutr. 2019 May 1;109(5):1328-1334. doi: 10.1093/ajcn/nqy390. PMID 31028699
- [Derived] Koppel N, Bisanz JE, Pandelia ME, Turnbaugh PJ, Balskus EP. Discovery and characterization of a prevalent human gut bacterial enzyme sufficient for the inactivation of a family of plant toxins. Elife. 2018 May 15;7:e33953. doi: 10.7554/eLife.33953. PMID 29761785
- [Derived] Hall KD, Chen KY, Guo J, Lam YY, Leibel RL, Mayer LE, Reitman ML, Rosenbaum M, Smith SR, Walsh BT, Ravussin E. Energy expenditure and body composition changes after an isocaloric ketogenic diet in overweight and obese men. Am J Clin Nutr. 2016 Aug;104(2):324-33. doi: 10.3945/ajcn.116.133561. Epub 2016 Jul 6. PMID 27385608
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0212.html